CLINICAL TRIAL: NCT05336786
Title: Prostate Cancer Diagnosis by Multiparametric Ultrasound (Wholemount)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Flemming Forsberg, Professor - Radiology, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21G.1212; R01CA252311 (NIH); JT 18100 (Other: JeffTrial Number)
Record Dates: First submitted 2022-04-07; First posted 2022-04-20 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — perflutren; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (perflutren lipid microspheres, ultrasound) (Experimental): Patients receive perflutren lipid microspheres IV over 5-6 minutes and undergo ultrasound over 30 minutes. Patients may receive up to 2 additional doses of perflutren lipid microspheres
  Interventions: Drug: Perflutren Lipid Microspheres; Procedure: Ultrasound

INTERVENTIONS:
Drug: Perflutren Lipid Microspheres — Given IV
  Other Names: Definity
Procedure: Ultrasound — Undergo ultrasound

SUMMARY:
This phase III trial investigates if perflutren lipid microspheres with ultrasound can be used to diagnose prostate cancer non-invasively. Definity (perflutren lipid microspheres) is an ultrasound contrast agent that is typically used for ultrasound bubble studies that involve the heart. Definity appears on ultrasound images as tiny gas-filled microbubbles. These microbubbles are about the size of a red blood cell and do not stay in a patient's body for more than several minutes, where they are excreted from the lungs and exhaled back into the air when breathing. Definity may enhance ultrasound images of the prostate and help doctors identify prostate cancer on ultrasound images.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect multiparametric ultrasound (mp-US) data on 70 patients within 30 days of their radical prostatectomy.

II. To correlate the imaging data with whole mount prostatectomy specimens in order to optimize mp-US with a machine learning approach.

OUTLINE:

Patients receive perflutren lipid microspheres intravenously (IV) over 5-6 minutes and undergo ultrasound over 30 minutes. Patients may receive up to 2 additional doses of perflutren lipid microspheres during ultrasound.

After completion of study, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be scheduled for radical prostatectomy for treatment of prostate cancer
* Subject must be able and willing to give written informed consent for a contrast enhanced ultrasound study of the prostate prior to prostatectomy
* Subject must be a male at least 18 years of age when informed consent is obtained

Exclusion Criteria:

* Participant in a clinical trial involving an investigational drug within the past 30 days
* Patients with known or suspected hypersensitivity to perflutren, PEG, or any other component of Definity
* Previous treatment for prostate cancer, including hormone therapy
* Clinically unstable, severely ill, or moribund as per treating physician

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Multiparametric ultrasound (mp-US) data to identify sites of significant malignancy within the prostate | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States
- Amsterdam University Medical Centers, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No